CLINICAL TRIAL: NCT05408221
Title: Phase Ⅱ/III Studies to Investigate the Efficacy and Safety of Rulonilimab in Combination With Lenvatinib Compared to Placebo in Combination With Lenvatinib as First-Line Therapy in Subjects With Hepatocellular Carcinoma
Brief Title: the Efficacy and Safety of Rulonilimab in Combination With Lenvatinib in Hepatocellular Carcinoma
Acronym: HCC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTP-F520-401
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rulonilimab (Experimental): with PD-1 Inhibitors
  Interventions: Drug: Rulonilimab+Lenvatinib
- Rulonilimab placebo (Placebo Comparator): without PD-1 Inhibitors
  Interventions: Drug: Rulonilimab placebo +Lenvatinib

INTERVENTIONS:
Drug: Rulonilimab+Lenvatinib — Rulonilimab, intravenous (i.v.) administration every 3 weeks; Lenvatinib oral administration, once daily
  Arms: Rulonilimab
Drug: Rulonilimab placebo +Lenvatinib — Rulonilimab placebo, intravenous (i.v.) administration every 3 weeks; Lenvatinib oral administration, once daily
  Arms: Rulonilimab placebo

SUMMARY:
There are two studies included in this protocol. One is an open-label Phase Ⅱ study . The other is a multi-center, double-blind, randomized, phase III study .

DETAILED DESCRIPTION:
There are two studies included in this protocol. One is an open-label Phase Ⅱ study designed to evaluate the tolerability and safety of lenvatinib in combination with Rulonilimab in participants with hepatocellular carcinoma (HCC). The other is a multi-center, double-blind, randomized, phase III study to investigate the efficacy and safety of Rulonilimab in combination with lenvatinib and placebo in combination with lenvatinib in the treatment of subjects with no prior systemic treatment and with unresectable advanced hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-75 full years (inclusive), male or female.
2. Subjects are with unresectable advanced HCC by histologically or cytologically confirmed diagnosis, Stage B or C based on Barcelona Clinic Liver Cancer [BCLC] ,that is not eligible for surgery and/or locoregional therapy or disease progression after surgery and/or locoregional therapy , surgery and/or locoregional therapy must be finished more than 4 weeks before baseline imaging scan .
3. Subjects have not received any systemic therapy for HCC previously (mainly including systemic chemotherapy, anti-angiogenic drugs or other molecular targeted therapy, antibodies/drugs targeting T cell co-regulatory proteins (such as anti-CTLA-4, anti-PD-1 /PD-L1, anti-OX-40, anti-CD137, anti-TIM-3, anti-LAG-3 antibodies, etc.).
4. Subjects with at least one measurable lesion by RECIST1.1, baseline imaging scan should be performed within 21 days prior to first administration，target lesions located in the field of previous radiotherapy or in the area of local treatment (interventional or ablative) are considered measurable if radiographic progression is confirmed.
5. Child-Pugh score A or B (≤7 ），There was no history of hepatic encephalopathy .
6. Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
7. Life expectancy ≥ 12 weeks.
8. The functions of vital organs meet the following requirements: No blood transfusion, no hematopoietic stimulating factors (including G-CSF, GM-CSF, EPO, TPO, etc.) and human albumin preparation are required within 14 days before the first administration:

   Blood test: neutrophil count (ANC) ≥1.5×109/L, hemoglobin (HGB) ≥90g/L, platelet count (PLT) ≥75×109/L; liver function: Total bilirubin level (TBIL) ≤2×ULN, ALT and AST≤5×ULN; kidney function: serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥50mL/min (Cr>1.5 x ULN); coagulation function: International standardized ratio (INR) ≤1.5×ULN; serum albumin ≥29g/L; urine protein <2+ (if urine protein ≥2+, 24h urine protein quantification should be performed, 24h urine protein quantification< 1.0g can be included).
9. Subjects with hepatitis B virus infection,and HBV DNA <2000 IU/mL during the screening period , willing to receive anti-HBV therapy throughout the study period.
10. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion criteria:

1. Fibrolamellar-HCC, sarcomatoid, cholangiocellular carcinoma or mixed cholangiocarcinoma and HCC.
2. History of other malignancy(ies) in the past 5 years, except for locally curable cancers (radical melanoma, basal or squamous cell carcinoma, carcinoma in situ of the bladder or cervix, etc.).
3. Palliative radiotherapy was performed for bone metastases within 2 weeks prior to firstl administration; Received drugs with anti-liver cancer effect (including Traditional Chinese medicine preparations) within 2 weeks before the first administration.Toxicity induced by previous therapy (except alopecia) not recovered to ≤ grade 1 (NCI-CTCAE v5.0).
4. Uncontrolled pericardial effusion, uncontrolled pleural effusion or clinically obvious moderate peritoneal effusion at screening.
5. Serious, uncured wound, active ulcer or untreated bone fracture.
6. History of gastrointestinal hemorrhage within 6 months prior to initial administration or clear tendency of gastrointestinal hemorrhage (including severe esophageal-gastric varices with hemorrhagic risk, locally active peptic ulcer, persistent fecal occult blood (+)).
7. Inability to swallow tablets, malabsorption syndrome or any other condition that affects gastrointestinal absorption.
8. Having ≥ grade 3 (NCI-CTCAE v5.0) gastrointestinal or non-gastrointestinal fistula at present.
9. According to CT/MRI examination, the main portal vein carcinoma thrombus involved the contralateral portal vein branch or the superior mesenteric vein at the same time;inferior vena cava carcinoma thrombus ;
10. Serious cardiovascular and cerebrovascular diseases:

    Appears New York Heart Association (NYHA) grade II or above congestive heart failure, unstable angina, myocardial infarction or cerebrovascular accident or poorly controlled arrhythmia within 12 months before the first administration (QTc interval ≥480ms, QTc interval calculated by Fridericia formula).

    LVEF (left ventricular ejection fraction) < 50%; uncontrolled hypertension (systolic blood pressure ≥150mmHg and/or diastolic blood pressure ≥100mmHg) (the average of ≥3 BP readings based on ≥2 measurements); has a hypertensive crisis or hypertensive encephalopathy.
11. Other obvious hemorrhagic tendency or evidence on important coagulation disorder:

    clinically significant hemoptysis or tumour hemorrhage of any cause within 4 weeks before first administration; a thrombosis or embolism event occurs within 6 months before first administration (e.g., aortic aneurysm or peripheral artery thrombosis requiring surgical repair; Uncontrolled deep vein thrombosis); use of anticoagulant therapy for therapeutic purposes (except low molecular weight heparin) within 2 weeks before first administration; requires antiplatelet therapy.
12. Medium or major surgery within 4 weeks prior to initial administration, but diagnostic biopsy was not included.
13. Central nervous system metastasis; If suspected, an MRI scan of the brain and/or spinal cord should be performed to rule it out.
14. For those who received live (attenuated) vaccines within 28 days prior to first administration or who planned to receive vaccines during the study period, the seasonal influenza vaccine for injection or COVID-19 vaccine is usually an inactivated virus vaccine and is allowed to be administered during the study period.
15. Presence of immunodeficiency or receiving long-term systemic steroid therapy within 7 days prior to randomization (daily dose >10mg Prednisone or other equivalent glucocorticoid), or other immunosuppressive therapy.
16. Active autoimmune diseases requiring systemic treatment (i.e., immunomodulatory drug, corticosteroid or immunosuppressant) in the past two years; Except for:

    alternative therapy (e.g. thyroxine, insulin or physiologic corticosteroid replacement therapy due to adrenal or pituitary insufficiency); a patient with well-controlled eczema, psoriasis, chronic simple moss or vitiligo with skin manifestations only, meeting the requirements of a rash ≤10% of body surface area and requiring no systemic drug therapy (including but not limited to hormones, immunosuppressants, etc.).
17. History of clear interstitial lung disease or non-infectious pneumonia, unless induced by local radiotherapy.
18. Active tuberculosis or received antituberculosis therapy within 1 year prior to randomization.
19. Any serious acute and chronic infection requiring systemic antibacterial, antifungal or antiviral therapy at screening, not including viral hepatitis.
20. A known history of human immunodeficiency virus (HIV) infection; Treponema pallidum antibody positive; HCV antibody positive and HCV-RNA positive or higher than the upper limit of normal value.
21. Previously receiving solid organ transplantation.
22. Known contraindication or history of hypersensitivity to any investigational drug or any known excipient.
23. Women who are pregnant or lactating, Female subjects at childbearing age or male subjects whose partners are of childbearing potential do not agree with contraception during the study period and for 6 months after the last administration.
24. Other participants who are unsuitable for inclusion as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
ORR | From randomization to PR or CR.Up to approximately 35 months.
  Objective Response Rate (ORR) Based on RECIST 1.1 Assessed by Independent Review Committee(IRC)

SECONDARY OUTCOMES:
PFS | From randomization to the first documented disease progression or death due to any cause, whichever occurs first.Up to approximately 35 months.
  Progression-free survival (PFS) evaluated by the Blinded Independent Central Review
OS | From date of randomization until the date of death from any cause.Up to approximately 35 months.
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Cai Jian qiang, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Zhou Ai ping, professor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (5):
- China (5):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Huizhou Central People's Hospital, Guandong
  - Jinan Central Hospital, Shandong
  - Linyi Cancer Hospital, Shandong
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen

IPD SHARING:
Plan to Share IPD: No